CLINICAL TRIAL: NCT05104151
Title: Evaluation of the Efficacy of a Nutritive Bar, in Reduction of Weight, Body Fat and Control of Appetite, in Patients With Overweight or Obesity in the City of medellín, 2017
Brief Title: Efficacy of a Nutritive Bar, in Reduction of Weight, Body Fat and Control of Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CES University (Other)
Responsible Party: Principal Investigator, Uriel Palacios, MD, CES University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 668
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Overweight or Obesity
Keywords: protein; weight control; appetite; overweight and obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: The proposed study is a randomized, single-blind, single center, parallel study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with nutritional bar (Experimental): Participants will recieve two nutritional bars per day during eight weeks, and will receive a healthy habits intervention wich includes: nutritional intervention providing a caloric deficit of 500 calories, and a prescription of moderate physical activity from 60 to 90 minutes daily.
  Interventions: Dietary Supplement: Nutritional bar; Behavioral: Healthy Habits Intervention
- Group without nutritional bar (Active Comparator): Participants will receive a healthy habits intervention wich includes nutritional intervention providing a caloric deficit of 500 calories, and a prescription of moderate physical activity from 60 to 90 minutes daily during eight weeks.
  Interventions: Behavioral: Healthy Habits Intervention

INTERVENTIONS:
Dietary Supplement: Nutritional bar — Protein-based nutritional bar, providing 155 calories per bar
  Arms: Group with nutritional bar
Behavioral: Healthy Habits Intervention — The participants included, will receive a nutritional intervention providing a caloric deficit of 500 calories, depending on their daily requirements, these daily requirements calculated according to the formula BMR (Basic Metabolic Rate). Also prescription of moderate physical activity from 60 to 90 minutes daily will be made.

SUMMARY:
The main objective of the trial is to measure the efficacy of a nutritive bar, in the reduction of weight, body fat and the control of appetite, in patients with overweight and obesity. It will be a randomized single-blind design conducted in 40 subjects.

DETAILED DESCRIPTION:
Primary objective and outcome: Difference in body fat percentage and summation of the absolute value of 7 body folds

Secondary objectives and outcomes:

* Characterize demographically and clinically the population participating in the research study.
* Determine the differences in body weight between the study groups.
* Determine the median of minutes of appetite onset in each of the groups. Design: The proposed study is a randomized, single-blind, paralell, single center study. Number of subjects: The number of subjects will be 40. At the start of the study, subjects will be randomly assigned to 2 different groups. All participants will have a evaluation with a nutritionist for an anthropometric assessment that includes the measurement of percentage of fat, sum of body folds, weight, height and Body Mass Index. All participants will receive a nutritional intervention providing a caloric deficit of 500 calories, depending on their daily requirements,and they will be prescribed moderate physical activity from 60 to 90 minutes daily. Participants will then be randomly assigned to gruop A: the nutritional bar group or group B: Control. Participants in group A will be instructed to consume the nutritional bar as an integral part of the previously established caloric regimen so as not to increase the number of prescribed calories and will be instructed to consume the product twice a day during the whole study, approximately 2 to 4 hours after breakfast and 2 to 4 hours after lunch, without additions of other foods or beverages, during consumption, may only be accompanied with water. Participants in group B will be instructed to consume a nutritious snack corresponding to the amount of calories provided by the bar, 2 to 4 hours after breakfast and 2 to 4 hours after lunch. The nutritional intervention will be carried out for 8 weeks for both groups, during the forth week and during the eight week of the intervention, a new nutritional assessment will be carried out with the same protocol of the first evaluation, by a nutritionist to all participants.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity (BMI range between 25.0 and 35 kg per m2 and
* Percentage of fat ≥28 for women and ≥20 for men

Exclusion Criteria:

* Pregnant
* People with gastrointestinal, thyroid, renal, hepatic or cardiovascular diseases.
* Diabetics or hypertensive.
* People with eating disorders.
* Use of anti-obesity drugs in the last 4 weeks.
* Use of nutritional or medicinal anti-obesity supplements in the last 4 weeks.
* Celiac Disease.
* Allergies to peanuts, nines, eggs, milk or products derived from milk.
* Vegans.
* Physical or mental disability.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2021-06-13 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Difference in body fat percentage | These measuremen will be made on: day one of study start for each particinat, during the fourth week of each participant of the study and during the eighth (last week) of the study for each participant
  The difference in changes of corporal body fat will be measured by calculating the percentage of body fat and the summation of the absolute value of 7 body folds. The percentage of body fat will be determined by using the Siri equation (% Fat = 4.95 / Dc) - 4.50 x 100), the calculation of the body density by the Jackson and Pollock anthropometric equation Dc = 1.10938 - 0.0008267 (sum of three folds) + 0.0000016 (sum of three folds) 2 - 0.0002574 years), the body folds for this outcome will be performed according to the International Society for the Advancement of Cineanthropometry (ISAK) protocol, with the body adipometer Harpenden (In women: Triceps, supraspinal and anterior thigh) (in men: pectoral, abdomen and thigh).

SECONDARY OUTCOMES:
Difference in body weight | This measuremen will be made on: day one of study start for each particinat, during the fourth week of each participant of the study and during the eighth (last week) of the study for each participant
  The subjects will be weighed by means of a balance SECA 813
Determine the median of minutes of appetite onset in each of the groups. | These levels will be measured over two days over the course of week one of the study for both groups
  The level of appetite after consumption of the food will be evaluated using an analogue visual scale (AVE). The AVE for appetite ranges from "0" (least appetite) to 10 (maximum appetite or hunger) and will be printed on sheets that will be delivered to the participants on the day of their nutritional evaluation and also by email, in case the lose Participants will be asked to either consume the product for group A or the isocaloric food recommended by the nutritionist for group B for two moments in the day (mid-morning or second feeding of the day and during the mid-afternoon or the fourth meal of the day), the subjects will be asked to write in the format the time of food intake, then the subjects must complete the EVA appetite scale every half hour for 2 hours. write by text message to the researchers the time of food consumption, so that they remind participants to fill out the form every 30 minutes.
Difference in summation of the absolute value of 7 body folds | This measuremen will be made on: day one of study start for each particinat, during the fourth week of each participant of the study and during the eighth (last week) of the study for each participant
  The body folds for this outcome will be performed according to the International Society for the Advancement of Cineanthropometry (ISAK) protocol, with the body adipometer Harpenden, the 7 body folds will be (triceps, biceps, subscapular, abdominal, supraspinal, anterior thigh and middle leg), and then will be made the summation of the absolute value of these 7 body folds

CONTACTS AND LOCATIONS:
Overall Officials: Uriel Palacios, MD, Principal Investigator — Professor
Locations (1):
- CES University, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Undecided
IPD will not be shared because the privacy of the participants will be guaranteed by not divulging their names in the scientific study process, or publication.